CLINICAL TRIAL: NCT02495480
Title: A Novel Disposable Sheathed Gastroscopic System for Cecal Intubation：Safety and Efficacy in Unsedated Colonoscopies
Brief Title: Disposable Sheathed Gastroscopic System for Cecal Intubation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yuqi He (Other)
Responsible Party: Sponsor-Investigator, Yuqi He, Doctor, General Hospital of Beijing PLA Military Region
Organization: General Hospital of Beijing PLA Military Region (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: GHBeijing
Record Dates: First submitted 2015-07-06; First posted 2015-07-13 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-07

CONDITIONS: Cecal Intubation Success Rate
Keywords: disposable sheath; intubation; colonoscopy

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- sheathed group (Experimental): The sterilized disposable sheath covered the outer surface of the colonoscope, then colonoscope will be performed in conventional way;a new sheath will be placed on the endoscope in sheathed group as a intervention
  Interventions: Device: A novel disposable sheath
- conventional group (No Intervention): Colonoscopy will be performed with air insufflation during insertion

INTERVENTIONS:
Device: A novel disposable sheath — a new sheath will be placed on the endoscope in sheathed group
  Arms: sheathed group

SUMMARY:
A novel disposable sheathed gastroscope system has been shown to be safe and more efficient in clinical practice during gastroscopy. This novel disposable sheathed endoscope system could effectively prevent cross-infection by simply taking off the contaminated sheath after examination of a patient and placing a new sheath on the endoscope. In this way, investigators can save the endoscopic reprocessing time and also decrease the need for endoscopic cleaning and disinfecting equipment.

Participants may think that placing a new sheath on the endoscope can decrease the success rate of cecal intubation in patients undergoing screening colonoscopy. With a new sheath on the endoscope during scope insertion can probably increases distension of the colonic lumen and loop formation. The probable adhesion may increase the discomfort of investigators and participants. But a previous clinical study by investigators' team showed that the participants' feeling were no significant difference (Z = -1.783, P = 0.075) between sheathed and conventional groups. No significant differences were observed in optical clarity, or pathology detection rate. There were no complications, and no microbial contamination was detected. Based on this study, investigators hypothesize that compared with conventional group, placing a new sheath on the endoscope does not significantly reduce the success rate of cecal intubation in average patients.

The aim of the study is to compare the outcome of colonoscopy placing a new sheath on the endoscope versus the conventional method in average participants. The primary outcome is cecal intubation success rate. The secondary outcomes include cecal intubation time, maximum pain score during colonoscopy, overall pain score after colonoscopy and adenoma detection rate.

ELIGIBILITY:
Inclusion Criteria:

* patients accepted sedated colonoscopy

Exclusion Criteria:

* a request for sedation/analgesia at the start of the procedure
* previous colorectal surgery
* declining to provide informed consent
* advanced comorbidity
* coagulopathy or anticoagulant medication administered
* failure to comply with the recommended bowel preparation regimen.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-07; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Cecal intubation success rate | up to ten months

SECONDARY OUTCOMES:
Pain according to a 10-point pain scale | up to ten months